CLINICAL TRIAL: NCT06851780
Title: Examining The Effect of Physical Workload on Postural Parameters in Physiotherapy and Rehabilitation Students
Brief Title: Analyzing Postural Parameters in Physiotherapy and Rehabilitation Students
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Asude ARIK, Research Assistant- PT, PhD, Hacettepe University
Other Study IDs: SBA 23/427
Record Dates: First submitted 2024-10-28; First posted 2025-02-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Health Risk Behaviors; Health-Related Behavior
Keywords: posture; work load; sleep quality; quality of life
MeSH Terms: conditions — Health Risk Behaviors; Health Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, with the voluntary participation of Term 3 and Term 4 students from the Hacettepe University Faculty of Physiotherapy and Rehabilitation, we examined the effect of physical workload on postural parameters based on students' standing and sitting times. Additionally, through surveys, we assessed the students' physical activity levels, quality of life, sleep, and burnout levels. The aim was to investigate the relationship between these components and postural alignment by measuring their levels. By identifying the factors that may affect students' postural alignment, the study aims to determine potential risks and provide valuable information for physiotherapists, physiotherapy students, and educators.

DETAILED DESCRIPTION:
Volunteer individuals among Term 4 (senior year) intern physiotherapist students and Term 3 students studying at Hacettepe University Faculty of Physical Therapy and Rehabilitation will be included in the study. Individuals who will be included in the study will be informed face to face about the purpose of the research, the evaluation methods to be used in the research, and the results we foresee, as well as what benefits we will provide to the individuals at the end of the study. Participants will be reached via posters/brochures. Individuals participating in the study will be informed about the surveys and the parameters to be evaluated at the first meeting. Postural evaluations of individuals will be carried out 4 times, on Mondays and Fridays, in the morning and in the evening, for 1 week. Questionnaires will be asked to be answered after the first and last posture evaluation. The number of individuals to be included in our study was calculated using the G*Power 3.1 program, taking the effect size as 0.74, alpha type error rate as 0.05 and the power of the test as 0.80, and the sample size for the period 4 and period 3 research groups was determined as 37/37. Taking into account situations such as inability to continue working, a total of 74 individuals were planned to be included in the study, with an excess of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study,
* Individuals who did not have pain according to the NORDIC Extended Musculoskeletal System questionnaire at the time of the evaluations,

Exclusion Criteria:

* Being diagnosed with scoliosis by a physician,
* Having spinal cord or extremity pain diagnosed by a physician in the last 3 months,
* Being diagnosed with any developmental disorder (Scheuermann's/Calve Disorder etc.),
* Having limb inequality, spine and pelvis etc. having serious deformities,
* Getting diagnosed with Infection (Spinal Tuberculosis etc.), Tumor (Multiple Myeloma),
* Having had spine surgery,
* Having a systemic inflammatory disease,
* Being diagnosed with a neurological and/or cognitive disease that may affect cognitive functions,
* Epilepsy, Antidepressant / Attention enhancing drug use,
* Being diagnosed with Cardiorespiratory Disease,
* Having menstrual irregularity,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Volunteer individuals from Term 4 (senior year) intern physiotherapist students and Term 3 students studying at Hacettepe University Faculty of Physical Therapy and Rehabilitation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2025-10-02 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Postural assessment | Up to four weeks
  Participants' postures will be evaluated using the Diers Formetric-4D system (DIERS International GmbH; Schlangenbad, Germany) operating with the Dicam 3v3.11 software. In this method, white light raster lines are projected onto the individual's back, and the deformation of these lines due to the 3D shape of the back is captured by a camera. The software detects convex and concave regions, allowing for the immediate identification of anatomical landmarks and fixed points. Using a mathematical algorithm, the system reconstructs a 3D model of the spine.During the measurement, participants will be positioned in a relaxed, motionless stance, standing on both feet, with their arms hanging freely, facing forward, and their backs turned toward the camera. Their heels will be placed on a marked area on the platform to ensure standard positioning.

SECONDARY OUTCOMES:
Musculoskeletal assessment | Baseline
  The Extended Nordic Musculoskeletal questionnarie will be used for the evaluation of musculoskeletal system. This questionnaire is used to identify musculoskeletal disorders and evaluates the body in nine regions: neck, shoulders, back, elbows, wrists/hands, lower back, hips/thighs, knees, and ankles/feet. It provides information on the onset, frequency, and consequences of musculoskeletal pain.
  The questionnaire first asks about the presence of pain or discomfort in these nine body regions. If the participant answers "yes", they proceed to the relevant follow-up questions.
  The Extended Nordic Musculoskeletal Questionnaire (NMQ-E) assesses whether pain, discomfort, or aches have been experienced at any time in life, in the past 12 months, in the past four weeks, and on the day of assessment.
Physical activity assessment | Baseline
  The International Physical Activity questionnaire will be used for the evaluation of physical activity. The short version of the International Physical Activity Questionnaire (IPAQ-SF) will be used to determine the type of physical activity an individual has performed in the past 7 days and the time spent on these activities. The total score will be calculated by multiplying the duration (minutes) and frequency (days) of walking, moderate, and vigorous activities.
  Participants will be classified based on their Metabolic Equivalent of Task (MET) score as follows:
  * Active: Above 3000 MET-min/week
  * Moderately active: Between 600 and 3000 MET-min/week
  * Inactive: Below 600 MET-min/week
Anxiety level assessment | Baseline
  The State-Trait Anxiety Inventory (STAI-1 and STAI-2) will be used for the evaluation of anxiety level. The STAI consists of 40 statements divided into two subscales: State Anxiety (STAI-1) and Trait Anxiety (STAI-2), each containing 20 items. It is a self-assessment questionnaire based on a 4-point Likert scale.
  * High scores (60-80) indicate high anxiety levels.
  * Moderate scores (40-59) indicate moderate anxiety levels.
  * Low scores (20-39) indicate low anxiety levels.
Sleep quality and disorder assessment | Baseline
  The Pittsburgh Sleep Quality Index will be used for the evaluation of sleep quality and disorder. The Pittsburgh Sleep Quality Index (PSQI) is a 24-item questionnaire designed to assess sleep quality and disturbances over the past month. Among these, 19 questions are self-reported, while 5 questions are answered by the spouse or roommate.
  Only 18 questions are scored, categorized into 7 components:
  1. Subjective Sleep Quality
  2. Sleep Latency
  3. Sleep Duration
  4. Habitual Sleep Efficiency
  5. Sleep Disturbances
  6. Use of Sleep Medication
  7. Daytime Dysfunction Each component is scored between 0 and 3, and the total score ranges from 0 to 21.
     * A total score above 5 indicates poor sleep quality.
     * A higher total score reflects worsening sleep quality.
Burnout level assessment | Baseline
  The malsach Burnout Inventory will be used for the evaluation of burnout level. The Maslach Burnout Inventory (MBI) is a 5-point Likert-type scale consisting of 22 items designed to assess occupational burnout. It is divided into three subscales:
  * Emotional Exhaustion (9 items)
  * Depersonalization (5 items)
  * Personal Accomplishment (8 items)
  Each item is scored on a scale from 0 to 4, where:
  * 0 = Never
  * 1 = A few times a year
  * 2 = A few times a month
  * 3 = A few times a week
  * 4 = Every day After scoring, each subscale's total score is calculated separately.
  * Higher scores in Emotional Exhaustion and Depersonalization indicate higher levels of burnout.
  * Higher scores in Personal Accomplishment indicate lower levels of burnout.
Quality Of Life Level assessment | Baseline
  The SF-36 Quality of Life Scale will be used for the evaluation of quality of life level. The Short Form-36 (SF-36) is a widely used self-reported health assessment questionnaire consisting of 36 questions across eight subscales: Physical Functioning, Role Limitations, Social Functioning, Mental Health, Vitality, Pain, and General Health. Each subscale is scored separately, and the total score ranges from 0 to 100. A higher score indicates a better health status and greater improvement in overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Gülce TANIMLI, Study Chair — Hacettepe University; Büşra ERGİT, Study Chair — Hacettepe University; Zafer ERDEN, Prof, Study Chair — Hacettepe University; Esra ATEŞ NUMANOĞLU, PhD, Study Chair — Hacettepe University; Asude ARIK, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degenhardt BF, Starks Z, Bhatia S. Reliability of the DIERS Formetric 4D Spine Shape Parameters in Adults without Postural Deformities. Biomed Res Int. 2020 Feb 13;2020:1796247. doi: 10.1155/2020/1796247. eCollection 2020. PMID 32104678
- [Background] Sorensen CJ, Norton BJ, Callaghan JP, Hwang CT, Van Dillen LR. Is lumbar lordosis related to low back pain development during prolonged standing? Man Ther. 2015 Aug;20(4):553-7. doi: 10.1016/j.math.2015.01.001. Epub 2015 Jan 14. PMID 25637464
- [Background] Poitras S, Blais R, Swaine B, Rossignol M. Management of work-related low back pain: a population-based survey of physical therapists. Phys Ther. 2005 Nov;85(11):1168-81. PMID 16253046
- [Background] Korakakis V, O'Sullivan K, O'Sullivan PB, Evagelinou V, Sotiralis Y, Sideris A, Sakellariou K, Karanasios S, Giakas G. Physiotherapist perceptions of optimal sitting and standing posture. Musculoskelet Sci Pract. 2019 Feb;39:24-31. doi: 10.1016/j.msksp.2018.11.004. Epub 2018 Nov 17. PMID 30469124
- [Background] Andersen JH, Haahr JP, Frost P. Risk factors for more severe regional musculoskeletal symptoms: a two-year prospective study of a general working population. Arthritis Rheum. 2007 Apr;56(4):1355-64. doi: 10.1002/art.22513. PMID 17393441